CLINICAL TRIAL: NCT00737802
Title: In Vivo Anatomy, Physiology, Mechanics and Function of the Lower Esophageal Sphincter
Status: Terminated | Type: Observational
Why Stopped: Was not able to recruit the total anticipated number of subjects
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Larry Miller, Principal Investigator, Northwell Health
Other Study IDs: R01DK059500 (NIH)
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: GERD; Barretts Esophagus
Keywords: GERD; Heartburn; Esophageal reflux; Barretts esophagus; Normal subjects
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus; Heartburn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal Control: Normal control subjects are the participants with no history of GERD, no signs and symptoms of GERD
- GERD Patients: GERD patients are those with history of GERD, signs and symptoms of GERD and selected signs and symptoms of GERD in the questionnaire.
- Barrett's patients: Barrett's patients are those participants who in addition to all the qualities of GERD patients have long standing history of GERD and mucosal changes in the esophagus.

SUMMARY:
The purpose of this study is:

* To study the components of the gastroesophageal junction high-pressure zone individually and as a group, by pharmacologically eliminating or accentuating the pressure profile generated by the smooth muscle components.
* To differentiate the gastric sling fibers from the clasp fibers based on the spatial orientation of these muscle groups.

DETAILED DESCRIPTION:
The purpose of this research study is to examine and evaluate a part of the digestive system (gastrointestinal tract). The specific part the study team will look at is called the "lower esophageal sphincter complex." This complex is located where the esophagus (food pipe) meets the top of the stomach. The lower esophageal sphincter complex involves a group of muscles, and the study team hopes to better understand how they work.

The study team hopes that, by studying the lower esophageal sphincter complex, it may be possible to discover how it functions and what causes it to fail. When a complex fails, this can lead to reflux and heartburn. So learning more about the lower esophageal complex may help doctors' better treat future patients with reflux problems.

We plan to study these functions in normal control subjects, in patients with GERD (heartburn symptoms), and in patients with Barrett's esophagus (a change in the lining of the esophagus due to chronic reflux). The doctor performing the study procedure has previous experience with and is skilled in performing these procedures.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for GERD patients are:

* Symptomatic heartburn
* Regurgitation
* Chest pain or water brash

Exclusion Criteria:

Exclusion criteria for normal volunteers include:

* Medications-Subjects on any medication which could effect the gastroesophageal junction high-pressure zone will be excluded, this includes use of antacids, H2 blockers, proton pump inhibitors, prokinetic agents, erythromycin type antibiotics and anticholinergics.
* GI symptoms, conditions and disorders

In addition exclusion criteria will include a history of:

* Esophagitis
* Gastrointestinal symptoms such as abdominal pain
* Heartburn
* Reflux
* Regurgitation
* Chest pain
* Difficulty swallowing
* Pain on swallowing
* Dysphagia
* Abdominal surgery involving the stomach or esophagus
* Nausea or vomiting
* Diabetes
* Scleroderma
* Esophageal motility disorders
* Non cardiac chest pain
* Achalasia and current pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal control subjects without GERD and patients with GERD
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2013-04-12 (Actual); Primary Completion 2015-04-09 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
Pressure at the gastric sling and clasp fibers | 5 years
  esophageal and gastroesophageal junction Pressure at the gastric sling and clasp fibers

CONTACTS AND LOCATIONS:
Overall Officials: Larry S Miller, MD, Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- LIJ Medical Center- NSLIJ Health System, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No